CLINICAL TRIAL: NCT07107087
Title: Multi-Modal Integrated Intervention Combining Exercise, Anti-inflammatory & Dietary Advice (MMIEAD) for Kidney Cachexia: a Mixed-methods Feasibility Cluster Randomised Controlled Trial and Process Evaluation
Brief Title: A Cluster Randomised Controlled Trial of a Multimodal Integrated Intervention for Kidney Cachexia
Acronym: MMIEAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Dr Joanne Reid, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B25/11
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Cachexia; CKD
MeSH Terms: conditions — Cachexia | interventions — Anti-Inflammatory Agents; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (MMIEAD + standard care) (Experimental): Individualised exercise programme:
  Participants will receive an exercise handbook and exercise diary to complete for a 12-week progressive home-based training programme (aerobic and resistance training). The intradialytic component will be an optional supervised 30-minute session up to 3 times per week.
  Dietary advice:
  Each patient in the intervention group will receive a 60-minute personalised dietetic assessment. Patients will be reviewed by the dietician at the start of the intervention and at 6-weeks and 12-weeks. Patients will also complete a 3-day food diary on five occasions throughout the 12 weeks of the interventions (weeks 1,3,6,9,12).
  Oral omega-3 supplement:
  Each patient will receive a 12-week supply of omega-3 oral capsules using a daily dose (1000mg twice daily) which has a proven safety profile, tolerability.
  Weekly contact:
  Patients in the intervention arm, will be contacted weekly (or more if preferred) by telephone. An adherence to MMIEAD log will be completed.
  Interventions: Other: Multi-Modal Integrated Intervention Combining Exercise, Anti-inflammatory & Dietary Advice (MMIEAD)
- Control arm (standard care) (No Intervention): Patients in the control arm will not be offered the MMIEAD intervention. All study sites have been surveyed to ensure the intervention components are not provided in standard care. Patients who have been allocated to the control group will be advised to adhere to routine standard care throughout the study. As the recruitment sites cover four Trusts, a description of standard care per Trust will be collected as part of the process evaluation.

INTERVENTIONS:
Other: Multi-Modal Integrated Intervention Combining Exercise, Anti-inflammatory & Dietary Advice (MMIEAD) — In addition to their standard care, the intervention group will receive MMIEAD - an individualised exercise programme, oral omega-3 supplementation and dietary advice.
  Arms: Intervention arm (MMIEAD + standard care)

SUMMARY:
This lay description has been written in conjunction with, and the content approved by our Patient and Public Involvement collaborators.

Patients with kidney cachexia will experience extreme muscle loss, reduced strength and symptoms including fatigue, reduced appetite and lower quality of life. Patients are also at an increased risk of hospitalisation and shortened life expectancy. Previous research suggests that treatments that target several causes of the muscle wasting syndrome (known as cachexia), show better outcomes for patients than treatments using just one method (for example only exercise). We want to see if combining different treatments (exercise, dietary advice and anti-inflammatory supplements) will improve outcomes for patients with kidney failure receiving haemodialysis at risk of developing kidney cachexia, compared to patients who only receive routine kidney care alone. However, there is currently no routine treatment for kidney cachexia. Individual treatments, such as exercise, have not been successful to slow the progression of wasting in chronic diseases. Our recent review of scientific literature highlighted dual treatments of exercise and dietary advice is effective to varying degrees. Combined treatments which include anti-inflammatory supplements (including those found in fish oils), alongside exercise and dietary advice, have been successfully trialled in other chronic illnesses, such as cancer for the treatment of cachexia. However, this bundle of three treatments has not been tested in patients with kidney cachexia. It is important to test whether such a combination of treatments will be practical for patients and clinicians. Our study will assess how well this intervention works in the healthcare system and if it shows potential to help patients with kidney cachexia.

Patients at risk of kidney cachexia who are receiving haemodialysis at two renal departments have been assigned to the treatment group (Multi-Modal Integrated intervention combining Exercise, Anti-inflammatory & Dietary advice plus routine care) and two have been assigned to the control group (routine care). Over 12 weeks, those in the treatment group will receive an individualised exercise programme, dietary advice and anti-inflammatory (fish oil) nutritional supplements. We will collect data on how successful the trial is (e.g., how many patients took part, completed all components of the study). Additionally, we will collect data on physical functioning, muscle mass, body weight, quality of life and survival. After 12 weeks, we will interview patients and clinicians to evaluate, if any, changes can be made to improve the intervention within what is called a 'process evaluation'.

ELIGIBILITY:
Inclusion Criteria:

* - CKD Stage 5 patients receiving maintenance HD therapy for >3 months, have oedema-free weight loss of at least 5% in 12 months or BMI less than 20 kg/m2, who have self-reported decreased physical function/muscle strength and appetite, increased fatigue, who are male or female, aged >18 years and able to provide written informed consent.

Exclusion Criteria:

* Patients under 18 years of age Patients within 3 months of initiation of HD (patients in this time frame are generally less clinically stable, many having vascular access procedures performed and with much higher rates of intercurrent events, including death and hospitalisation).

Patients experiencing weight loss due to clinically explainable reasons for example malabsorption or oesophageal blockage.

Patients already receiving chronic anticoagulation therapy or with a history of bleeding with 3 months/active bleeding issues.

Patients receiving immunosuppressants or immunomodulators. Patients who are pregnant or breast feeding. Patients with a hypersensitivity to any of the constituent components of the omega-3 dietary supplement Patients who have dementia, a psychiatric disorder (who are not treated and stable) or a severe cognitive impairment which would deem them unable to give informed consent.

Patients with expected survival on dialysis of <6 months [e.g. those with severe heart failure (New York Heart Association ≥3)].

Patients for whom dialysis withdrawal is being considered. Patients likely to receive a live-donor transplant or transfer to peritoneal dialysis during the study duration.

Patients with bilateral lower limb amputations. Patients unable to walk without aids or assistance. Patients deemed to be clinically unstable by their treating physician. Patients who are non-English speaking (not having the ability to provide informed consent, read and write English).

Patients who are currently enrolled in any study which involves exercise, fish oil/omega-3 or have been taking fish oil or omega-3 supplementation in the previous 3 months.

Are not able/willing to be involved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment; measured as the number of fully enrolled patients as a proportion of approached eligible individuals | From enrollment to the end of treatment at 12 weeks